CLINICAL TRIAL: NCT00124852
Title: The Efficacy of Omega-3 Fatty Acids in Maintaining Optimal Mental Health in Elderly People: a Double-blind Placebo-controlled Trial
Brief Title: The Efficacy of Omega-3 Fatty Acids in Maintaining Optimal Mental Health in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Prof Dr Lisette CPGM de Groot, Wageningen University
Organization: Wageningen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2005_05/08; 6100.0004
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Cognitive Impairment; Depression
Keywords: cognition; depression; elderly
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Oleic Sunflower Oil (Placebo Comparator)
  Interventions: Behavioral: n-3 Fatty Acid Supplementation
- 400 mg EPA+DHA/day (Active Comparator): low dose fish oil
  Interventions: Behavioral: n-3 Fatty Acid Supplementation
- 1800 mg EPA+DHA/day (Active Comparator): high dose fish oil
  Interventions: Behavioral: n-3 Fatty Acid Supplementation

INTERVENTIONS:
Behavioral: n-3 Fatty Acid Supplementation

SUMMARY:
The efficacy of EPA-DHA supplementation will be assessed in a randomized placebo-controlled trial with cognitive decline and early signs of depression as primary outcome measures.

DETAILED DESCRIPTION:
The efficacy of EPA-DHA supplementation will be assessed in a randomized placebo-controlled trial with cognitive decline and early signs of depression as primary outcome measures. In this study 300 elderly people will be randomly allocated to one of three treatments. Two groups will receive fish oil capsules with different doses EPA/DHA (a normal dose or a high dose) and the third group will receive placebo capsules. At the start and at the end of the intervention period cognitive function, the occurrence of depression, quality of life, anthropometric values and biochemical indicators will be measured.

After completion of the trial a workshop will be organized in which the outcomes of the proposed study will be presented to representatives of several key areas concerning mental health of elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 65 years and over
* Informed consent signed

Exclusion Criteria:

* A score of > 16 on the CES-D (Centre for Epidemiological Studies-Depression Scale
* A score of < 21 points on MMSE (Mini-Mental State Examination)
* Current or recent (<4 weeks) use of fish oil supplements or intake of more than 4 times fish as judged by a fish consumption questionnaire
* Current use of pharmacological antidepressants
* Current use of dementia (Alzheimer) medication
* Serious liver disease
* Use of more than 4 glasses of alcohol per day
* Unable to participate as judged by the responsible medical physician
* Allergy to fish(oil)
* Swallowing problems
* Participation in another clinical trial less than 2 months before the start of the trial or at the same time

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 302 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Cognitive function
Depression

SECONDARY OUTCOMES:
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Dr Ir, Study Director — Project leader; Marianne Geleijnse, Dr, Study Director — Project leader
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Bouwens M, van de Rest O, Dellschaft N, Bromhaar MG, de Groot LC, Geleijnse JM, Muller M, Afman LA. Fish-oil supplementation induces antiinflammatory gene expression profiles in human blood mononuclear cells. Am J Clin Nutr. 2009 Aug;90(2):415-24. doi: 10.3945/ajcn.2009.27680. Epub 2009 Jun 10. PMID 19515734
- [Derived] van de Rest O, Geleijnse JM, Kok FJ, van Staveren WA, Hoefnagels WH, Beekman AT, de Groot LC. Effect of fish-oil supplementation on mental well-being in older subjects: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2008 Sep;88(3):706-13. doi: 10.1093/ajcn/88.3.706. PMID 18779287